CLINICAL TRIAL: NCT00685607
Title: A Placebo-Controlled, Double-Blind, Randomized Pilot Study to Evaluate the Appropriateness of Multiple Endpoints in Measuring the Onset of Clinical Efficacy of Loperamide-Simethicone Caplets in the Treatment of Acute Non-specific Diarrhea
Brief Title: Study to Determine the Best Way to Measure How Quickly the Drug Can Give Relief From Sudden Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOPDIR4003
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Diarrhea
Keywords: Pilot Study; Outcome Measures
MeSH Terms: conditions — Diarrhea | interventions — Loperamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): loperamide-simethicone
  Interventions: Drug: loperamide-simethicone
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: loperamide-simethicone — Four caplets containing 2 mg loperamide HCl and 125 mg of simethicone each, administered orally with 4-8 oz. of water according to the labeled directions of the currently marketed product (i.e., 2 caplets after first loose stool, followed by 1 caplet after each subsequent loose stool, not to exceed 4 caplets in 24 hours). The treatment period will last six hours.
  Other Names: Imodium
  Arms: 1
Drug: matching placebo — Four placebo caplets matching the caplets in Arm 1, administered orally with 4-8 oz. of water according to the labeled directions of the currently marketed product (i.e., 2 caplets after first loose stool, followed by 1 caplet after each subsequent loose stool, not to exceed 4 caplets in 24 hours). The treatment period will last six hours.
  Other Names: Placebo
  Arms: 2

SUMMARY:
For six hours following drug administration, subjects will rate the severity of specific symptoms. At the end of the six hour study, subjects will rate the overall effectiveness of the product.

DETAILED DESCRIPTION:
A six-hour study to evaluate multiple early efficacy endpoints in loperamide-simethicone therapy to help identify speed of onset of symptomatic treatment of acute nonspecific diarrhea (ANSD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute diarrhea with gas-related abdominal discomfort, meeting specific criteria
* Willing to follow the protocol requirements and comply with protocol restrictions, including use of contraception
* Able to understand the informed consent process and sign the form
* Cooperative, reliable and willing to comply with the protocol requirements and schedule, and able to record efficacy and safety assessments.

Exclusion Criteria:

* Female subjects who are pregnant, lactating or experiencing perimenstrual abdominal or pelvic discomfort
* Illness requires hospitalization, IV fluids or antibiotics
* Has taken antibiotics in the past 7 days or a symptomatic antidiarrheal compound in the past 12 hours or any analgesic in the past 6 hours
* History of significant underlying enteric, pulmonary, hepatic, cardiac, renal disease, seizure disorder, IBD, cancer, uncontrolled diabetes, or any other unstable medical condition
* History of hypersensitivity to loperamide or simethicone
* Has previously participated in this study or received an investigational drug within the 30 day period before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evaluate Multiple Endpoints | 6 hours

SECONDARY OUTCOMES:
Time to improvement in stool form | 6 hours
Time to improvement in urge to defecate | 6 hours
Time to improvement in gas-related abdominal discomfort | 6 hours
Time to improvement of change in normal activities of daily living | 6 hours
Subject global impression of efficacy of study medication at the end of the treatment period | 6 hours
Physical examination and vital signs at the screening visit and the monitoring of adverse events throughout the course of the study | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L DuPont, MD, Study Chair — Department of Public Health, University of Texas, Houston School of Public Health
Locations (1):
- Universidad Autonoma de Guadalajara, Guadalajara, Jalisco, Mexico